CLINICAL TRIAL: NCT03476720
Title: Accuracy of Instructional Diagrams for Automated External Defibrillator (AED) Pad Positioning
Brief Title: Improving Defibrillation Pad Position
Status: Completed | Type: Observational
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: TBC
Record Dates: First submitted 2018-03-15; First posted 2018-03-26 (Actual); Last update posted 2018-10-22 (Actual); Status verified 2018-10

CONDITIONS: Cardiac Arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Pad positioning according to a manufacturer's diagram — Placement of defibrillation pads according to the diagram

SUMMARY:
Manufacturer's diagrams showing defibrillation pad positioning (as used on public access defibrillators) are anatomically incorrect and are likely to lead to poor position of defibrillation pads, with reduced defibrillation efficacy.

We will ask untrained members of the public to observe the diagrams and place pads as indicated on the diagram. We will asses the accuracy of pad placement and repeat the study using an anatomically correct diagram to see if we can improve the accuracy of pad placement.

DETAILED DESCRIPTION:
As above

ELIGIBILITY:
Inclusion Criteria:

- 16 yrs age and willing to participate.

Exclusion Criteria:

* Previous BLS training
* Previous AED training
* Clinical staff (doctor, nurse, HCA, paramedic etc)

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All adults who have had no training in basic life support or public access/AED defibrillation.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-04 (Actual)

PRIMARY OUTCOMES:
Pad position | 6 months
  Position of the pad (vertical and horizontal) in relation to optimal position as recommended by the resuscitation guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Deakin, MD, Study Director — University Hospital Southampton NHS Foundation Trust
Locations (1):
- University Hospital Southampton, Southampton, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No